CLINICAL TRIAL: NCT01859611
Title: Clinical Study to Evaluate the Performance of TriActive+ RF for the Non-Invasive Treatment of Wrinkles and Rhytides
Brief Title: TriActive+ Radiofrequency (RF) for Non-Invasive Treatment of Wrinkles and Rhytides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: El. En. SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TriActive+RF-ElEn-022013
Record Dates: First submitted 2013-05-10; First posted 2013-05-22 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Wrinkles; Rhytides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiofrequency (Experimental): Radiofrequency (RF) treatment with the TriActive+ RF device on the peri-oral and/or peri-orbital areas of the face once a week for eight weeks.
  Interventions: Device: TriActive+ RF

INTERVENTIONS:
Device: TriActive+ RF — Radio frequency handpiece uses a multi-polar technology with a particular electrical frequency of 1MHz. The handpiece has a special "skin contact identification" system which delivers energy only when electrodes are adherent to the skin surface in order to avoid the prickling sensation when the treatment starts.

SUMMARY:
The study objective is to evaluate the safety and efficacy of a radiofrequency (RF) source, the TriActive+ RF handpiece, for treatment of wrinkles and rhytides after multiple treatments. The primary endpoint is observation of changes to the surface by visual and photographic analysis. Secondary endpoints: measurement of patient satisfaction and comfort of the treatment and the measurement of adverse events.

DETAILED DESCRIPTION:
Collagen varies genetically and structurally. Collagen breakdown increases with chronological age and photoaging. While fibroblasts normally replace damaged collagen fibers with new ones, the ability of fibroblasts to replace collagen is compromised by natural aging and environmental stress. Although collagen fibers form a loose interlacing network that is deformable, increased collagen breakdown leads to thinning and loss of the elastic fiber network in the dermis. This breakdown results in the formation of wrinkles, especially in areas of the skin exposed to the sun, which are most prone to wrinkles and imperfections. Nonablative dermal remodeling has gained tremendous popularity among patients and practitioners, offering a low incidence of adverse effects and modest improvement in the various signs of cutaneous photoaging, including rhytides, dyschromias and telangiectasias. Controlled thermal skin injury has been shown to effect a conformational change in the structure and length of collagen and may also induce fibroblast response for long-term collagen remodeling. Interest in utilizing radiofrequency energy to enhance deep tissue tightening and thus improve skin laxity has grown, as radiofrequency energy has been shown in multiple studies to tighten tissue, producing a noticeable skin lifting.

This study is intended to evaluate the clinical performance of a radiofrequency (RF) source as engendered in the TriActive+ RF for the non-invasive treatment of wrinkles and rhytides.

Eligible subjects who have signed an ICF will receive up to 8 treatments on at least two facial sub areas (left peri-orbital, right peri-orbital and peri-oral). Up to 25 subjects will be enrolled in the study at two sites. Treatments will start at a low power and then gradually increase, based on tolerability and tissue reaction. The goal is to progressively reach and maintain an epidermal temperature end-point. The site will use an IR thermometer to ensure the rise in temperature does not exceed 43° C.

Treatments will be once a week with follow-up visits at one week, one month, and three months following the final treatment. Clinical assessments by the investigator and digital photographs will be taken prior to the baseline treatment, immediately prior to the 5th treatment, and at the 1 week, 1 month and 3 month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* ICA signed by the subject.
* Healthy male or female subjects 30-60 ys of age.
* Having at least 2 facial sub-areas (left peri-orbital, right peri-orbital or peri-oral) with visible lines/wrinkles and elastosis, which correlate to a score of 2-6 on the Fitzpatrick Classification of Wrinkling and Degree of Elastosis.
* Willingness to follow the treat and FU schedule and the post-treat care.
* For female candidates - post-menopausal or surgically sterilized or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire study

Exclusion Criteria:

* Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breastfeeding. Females of childbearing potential must agree to take a urine pregnancy test (must be negative) at the Screening visit. Females of childbearing potential include anyone who has experienced menarche and who has not undergone successful surgical sterilization or is not post-menopausal for more than 2 years.
* Having any active electrical implant anywhere in the body
* Having a permanent implant in the treated area or an injected chemical substance.
* Having a history of diseases stimulated by heat unless treatment is conducted following a prophylactic regimen.
* Use of non-steroidal anti-inflammatory drugs one week before and after each treatment session.
* Use of retinoids, antioxidants or skin nourishing supplements within 1 month of treatment or during the study.
* Having received a facial dermabrasion or chemical peel treatment within 2 months of treatment or during the study.
* Having received treatment with light, RF or other devices in the treated area within 6 months of treatment or during the study.
* Having received Botox in the treated area within 6 months or collagen/Hyaluronic Acid within a year of treatment or during the study.
* Having undergone a resurfacing procedure, face lift or eyelid surgery within a year of treatment or during the study.
* Having undergone any other surgery in the treated area within 6 months of treatment (or more if skin has not healed completely) or during the study.
* Having ever received fat injections or other methods of augmentation with injected or implanted material in the treated area or planning to during the study.
* History of keloid scarring or of abnormal wound healing.
* Suffering from current or history of significant skin conditions in the treated area or inflammatory skin conditions prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
* History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
* History of epidermal or dermal disorders.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Suffering from hormonal imbalance, as per the Investigator's discretion.
* Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course.
* Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
* Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), or pertinent neurological disorders.
* Vascular lesion, tattoo or permanent make-up in the treated area.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Participation in a study of another device or drug within 1 month prior to enrollment or during the study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Bizzari, ElEn, Study Director — El. En. SpA
Locations (2):
- United States (2):
  - Chernoff Plastic Surgery & Laser Center, Indianapolis, Indiana
  - Park Avenue SmartLipo, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period from April 2013 to August 2013 at two private offices
Period: Overall Study
Arm/Group | Radiofrequency
Started | 51
Completed | 43
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Changes to the Surface by Visual and Photographic Analysis.
Description: At each of the specified time points, photographs of the treated areas will be taken. The photography angles will include a global frontal photo and the right and left sides of the face at 45° and/or 90°. In addition, close up photos will be taken of specific facial zones, e.g., the peri-orbital wrinkles.
  Each patient to be evaluated through the 9 grade Fitzpatrick Wrinkling Severity Scale.
  Wrinkling Score Degree of Elastosis Fine 1-3 Mild Fine to moderate 4-6 Moderate Fine to deep wrinkles 7-9 Severe
Time Frame: 3 Month FU
Population: Number of participants with observed changes (grade of improvement ≥ 1) to the surface of the skin based on photographic analysis at 3 Month FU
Measure: Number; unit: participants
Arm/Group | Radiofrequency
Number analyzed (Participants) | 51
participants | 41

2. Secondary Outcome: Patient Satisfaction and Comfort of the Treatment.
Description: At each of the specified time points, subjects will complete a Subject Evaluation Form assessing their opinion of improvement and overall satisfaction with treatment.
Time Frame: Pre Treatment 5, 1 Week FU, 1 Month FU, 3 Month FU
Reporting Status: Not Posted

3. Secondary Outcome: Adverse Events.
Description: At every treatment and follow-up visit the treated areas will be examined to evaluate side effects and adverse reactions remaining from the previous treatment session or occurring since then.
Time Frame: Subjects will be followed for the duration of the study, and expected average of 20 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From May 2013 to January 2014
Arm/Group | Radiofrequency
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No